CLINICAL TRIAL: NCT05326061
Title: Characterization of Patients at High Risk for the Acquisition of Sexually Transmitted Infection With the Human Immunodeficiency Virus (HIV) - a Clinical Study
Brief Title: Vienna HIV Infection Via Sex Study
Acronym: HIVEX
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Armin Rieger, MD, Ass.-Prof. Dr.med.univ., Medical University of Vienna
Other Study IDs: 1051_2020
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: HIV Infections; HIV Pre-Exposure Prophylaxis; Sexually Transmitted Diseases; Gonorrhea; Chlamydia; Syphilis
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Gonorrhea; Chlamydia Infections; Syphilis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this prospective observational cohort study is to investigate the epidemiology, the risk factors and ultimately the incidence of novel HIV infections among individuals at high risk for acquiring HIV via sex practices.

DETAILED DESCRIPTION:
We will include individuals at high-risk for HIV acquisition, i.e. HIV-negative MSM and transgender individuals who (i) do not use condoms consistently with casual partners and/or with HIV-positive partners who are not on treatment and/or (ii) recently acquired an STI and/or (iii) recently used PEP and/or (iv) frequently engage in 'chemsex' within the past 12 months Important clinical information on possible vectors for transmission (including but not limited to high-risk sex practices and sexualized drug use), use of HIV pre-exposure prophylaxis, incidence of sexually transmitted infections will be assessed and laboratory parameters will be obtained from blood, urine and mucosal secretion.

ELIGIBILITY:
Inclusion Criteria:

1. High risk for acquiring HIV defined as followed: HIV-negative MSM and transgender individuals who (i) do not use condoms consistently with casual partners and/or with HIV-positive partners who are not on treatment and/or (ii) recently acquired an STI and/or (iii) recently used PEP and/or (iv) frequently engage in 'chemsex'.
2. Age >18 years and <100 years.
3. Written informed consent for this registry study.

Exclusion Criteria:

1. Withdrawal of the written informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting at the HIV- and/or STI ward of the Department of Dermatology at General Hospital of Vienna which are characterized as individuals at high risk for acquiring HIV will be considered as potential participants for the HIVEX registry.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of HIV | Up to 10 years (=Study Period)
  Time from inclusion to HIV infection

SECONDARY OUTCOMES:
Incidence of sexually transmitted infections | Up to 10 years (=Study Period)
  Time from inclusion to any sexually transmitted infections

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria